CLINICAL TRIAL: NCT05829473
Title: The Effect of Guided Imagery and Diaphragmatic Breathing Exercise on the Severity of Nausea, Vomiting and Anxiety Level in Pregnants With Hyperemesis Gravidarum
Brief Title: The Effect of Guided Imagery and Diaphragmatic Breathing Exercise in Pregnant Women With Hyperemesis Gravidarum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hyperemesis Gravidarum
Record Dates: First submitted 2022-11-28; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Hyperemesis Gravidarum
Keywords: Anxiety; Hyperemesis Gravidarum; Nausea-Vomiting; Guided Imagery; Diaphragmatic Breathing Exercise
MeSH Terms: conditions — Hyperemesis Gravidarum; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breathing Exercise Group (Experimental): A total of 1 times day diaphragmatic breathing exercise will be made on 3 consecutive days (5 minutes diaphragmatic breathing exercise, 5 minutes relaxation exercise). Diaphragmatic breathing exercises will be performed at least 4 hours after the use of antiemetic drugs in the service. 20 minutes from the diaphragmatic breathing exercise application. Afterward, post-test data will be obtained using the Nausea-Vomiting Severity Evaluation Test During Pregnancy and Pregnancy-Related Anxiety scales. A total of 6 measurements will be made using the scales on the 1st, 2nd, and 3rd days.
  Interventions: Other: Breathing Exercise Group
- Guided Imagery Group (Experimental): 10 minutes once a day for pregnant women with hyperemesis gravidarum who meet the research criteria the guided imagery compact disc will be played with the computer. A guided imagery compact disc will be watched at least 4 hours after the use of antiemetic drugs in the service.10 minutes once a day for pregnant women with hyperemesis gravidarum who meet the research criteria the guided imagery compact disc will be played with the computer. A guided imagery compact disc will be watched at least 4 hours after the use of antiemetic drugs in the service. Afterward, 20 minutes from the application post-test data will be obtained by using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales. A total of 6 measurements will be made using the scales on the 1st, 2nd, and 3rd days.
  Interventions: Other: Guided Imagery Group
- Control Group (No Intervention): No intervention will be made to the pregnant women in the control group, other than their routine daily care. Pre-test data will be obtained by applying the Nausea-Vomiting Severity Evaluation Test During Pregnancy and Pregnancy-Related Anxiety scales at least 4 hours after the use of antiemetic drugs in the service. 20 min from the pre-test data. Afterward, the final test data will be obtained by applying the Nausea-Vomiting Severity Evaluation Test During Pregnancy and Pregnancy-Related Anxiety scales. A total of 6 measurements will be made using the scales on the 1st, 2nd, and 3rd days.

INTERVENTIONS:
Other: Breathing Exercise Group — A total of 1 times day diaphragmatic breathing exercise will be made on 3 consecutive days (5 minutes diaphragmatic breathing exercise, 5 minutes relaxation exercise). Diaphragmatic breathing exercises will be performed at least 4 hours after the use of antiemetic drugs in the service. 20 minutes from the diaphragmatic breathing exercise application. Afterward, post-test data will be obtained using the Nausea-Vomiting Severity Evaluation Test During Pregnancy and Pregnancy-Related Anxiety scales. A total of 6 measurements will be made using the scales on the 1st, 2nd, and 3rd days.
  Arms: Breathing Exercise Group
Other: Guided Imagery Group — 10 minutes once a day for pregnant women with hyperemesis gravidarum who meet the research criteria the guided imagery compact disc will be played with the computer. A guided imagery compact disc will be watched at least 4 hours after the use of antiemetic drugs in the service.10 minutes once a day for pregnant women with hyperemesis gravidarum who meet the research criteria the guided imagery compact disc will be played with the computer. A guided imagery compact disc will be watched at least 4 hours after the use of antiemetic drugs in the service. Afterward, 20 minutes from the application post-test data will be obtained by using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales. A total of 6 measurements will be made using the scales on the 1st, 2nd, and 3rd days.
  Arms: Guided Imagery Group

SUMMARY:
Objective: The aim of the researchers is to determine the effects of guided imagery and diaphragmatic breathing exercise application on nausea, vomiting severity, and anxiety level in pregnant with hyperemesis gravidarum.

Methods: This study was planned as a single-blind randomized controlled experimental study. It is planned to be conducted with 180 pregnant women to be randomized in a university hospital in Southeastern Anatolia between April 2023 and August 2023. Data will be collected using the "Descriptive Information Form", "Nausea-Vomiting Severity Assessment Test During Pregnancy" and "Pregnancy-Related Anxiety Scale-R2".

Keywords: Anxiety, Hyperemesis Gravidarum, Nausea-Vomiting, Guided Imagery, Diaphragmatic Breathing Exercise, Nursing,

DETAILED DESCRIPTION:
1. INTRODUCTION AND OBJECTIVE Pregnancy-related nausea and vomiting are attacks that occur in the first half of pregnancy, accompanied by occasional nausea and vomiting. Hyperemesis gravidarum is a clinical picture of unknown etiology and without standardization in its diagnosis and treatment. Hyperemesis gravidarum, on the other hand, although not a universally accepted definition, can generally be defined as a condition that causes a loss of 5% of the pre-pregnancy weight before the 20th gestational week, with vomiting severe enough to require hospitalization. It usually begins in early pregnancy (at 4-8 weeks) and lasts until the start of the second trimester. Hyperemesis gravidarum is seen in approximately 0.3-2% of pregnancies and is one of the most common causes of hospital admission in the first half of pregnancy.

   In the treatment of hyperemesis gravidarum, there are many non-pharmacological treatment methods as well as pharmacological methods. Alternatively, some non-pharmacological applications can be used alone or in combination with drug therapy as an adjunctive treatment option to control nausea and vomiting. These non-pharmacological methods; diet, music therapy, daydreaming, and hypnosis. In addition to these applications, there are also applications such as social support groups, regular exercise, vitamin drugs, aromatherapy, yoga, ginger root tea, breathing exercises, acupuncture, and reflexology/foot massage in controlling nausea and vomiting. Among these alternatives, non-pharmacological treatment methods are breathing exercises and guided imagery. There are studies showing that guided imagery and breathing exercise practices reduce stress and anxiety in pregnant women, increase their well-being, are beneficial to their daily lives, positively contribute to mother-baby bonding, and reduce pain in high-risk pregnant women.

   However, as a result of the literature review, it was seen that there was no study investigating the effects of guided imagery and diaphragmatic breathing exercise on the severity of nausea, vomiting, and anxiety level in pregnant women with hyperemesis gravidarum. Therefore, the aim of the researchers is to determine the effects of guided imagery and diaphragmatic breathing exercise application on nausea, vomiting severity, and anxiety level in pregnant with hyperemesis gravidarum.

   HYPOTHESES

   The hypotheses of this study are:

   H0: Diaphragmatic breathing exercises and guided imagery have no effect on nausea, vomiting severity, and anxiety level in pregnant with hyperemesis gravidarum.

   H1: Diaphragmatic breathing exercise reduces nausea and vomiting severity. H2: Diaphragmatic breathing exercise reduces anxiety level. H3: Guided imagery reduces nausea, vomiting severity H4: Guided imagery reduces anxiety levels.
2. MATERIAL AND METHODS 2.1. Study Design: This study was planned as a single-blind randomized controlled experimental study.

2.2. Setting and Samples: The researchers planned to be done this study between December 2022 and December 2023 in the gynecology and obstetrics service, at the university hospital in southeastern Anatolia, Turkey.

The sample size was assessed using G-power analysis (effect size 0.3; medium level α = 0.05; 1-β = 0.80), and it was found that for each group, 58 patients had the capability of representing the population. However, we decided to include 60 pregnant women in each group in order to be able to generalize and strengthen the research results.

2.2.1. Randomization: Medical version 18.11.3 will be used for the randomization list for assigning participants to groups. Pregnant women participating in the study won't know how many groups are available and which method will be applied to the group in which they are selected. We will do this study with three groups, two experiments, and one control. The experimental group will be divided into two groups, guided imagery, and breathing exercise group.

2.3. Data Collection Tools: The data of the study will be collected by using ''The Descriptive Information Form", "Nausea-Vomiting Severity Evaluation Test During Pregnancy ", and "Pregnancy-Related Anxiety Scale- R2 ''.

2.3.1. The Descriptive Information Form: This form, which was developed by researchers through a literature review, consists of three parts. In the first part, the age, education, duration of the marriage, income status, etc. of pregnant women. 10 questions, including socio-demographic characteristics such as; the second part includes the first gestational age, the number of miscarriages, gestational week, expected delivery date, etc. including obstetric features such as 7 questions; The third part consists of 2 questions evaluating the satisfaction with the applications made to the intervention groups. The introductory information form will be filled in by the researchers by communicating face-to-face on the first day of hospitalization to the intervention and control groups.

2.3.2. Nausea-Vomiting Severity Evaluation Test During Pregnancy: The scale consists of 3 questions questioning nausea, vomiting, and retching, respectively. Although the symptoms were initially questioned for the last 12 hours, it was later updated to cover the last 24 hours. When evaluating the Nausea-Vomiting Severity Evaluation test, the total score is stated as mild if it is 3-6, moderate if 7-12, and severe nausea and vomiting if it is 13-15.

2.3.3. Pregnancy-Related Anxiety Scale- R2: It is a 5-point Likert scale. The 11-item scale consists of "fear of childbirth (1, 2, 6, and 8th items)", "fear of having a disabled child (4, 9, 10, and 11th)" and "concerns about physical appearance (3, 5 and 7). item)" has 3 sub-dimensions. The 8th item in the scale (I am worried about childbirth because I have never given birth before) is used for women who have not given birth before but is not applied to multiparous women. Items are scored between 1-5 (1-Strongly disagree and 5-Strongly agree) and a minimum of 11 points and a maximum of 55 points are received for primiparas, and a minimum of 10 and a maximum of 50 points are received for multiparas. As the score obtained from the scale increases, it is accepted that the level of anxiety in pregnancy is higher. All of the expressions in the scale are positive. The scale has no cut-off point. The Cronbach's alpha coefficient of the scale was 0.93 for the multiparous group and 0.94 for the primiparous group.

2.4. Data Collection: After the approval of the ethics committee and the application permission of the research, the hospital head physician, head nurse, gynecology service physicians, and nurses will be interviewed and information will be given about the purpose and scope of the research. Data will be collected by the researcher. Pregnant women who comply with the sampling selection criteria and agree to participate in the study will be informed about the purpose of the research, the method of the research, the breathing exercise and guided imagery method in accordance with the group they belong to, and the hospital management and ethics in order to carry out the research, It will be explained that permission has been obtained from the committee, that identity information is required for research consent, that identity information will be kept confidential by the researcher, and their consent will be obtained with a verbal and Informed Voluntary Consent Form.

Breathing Exercise Group: An introductory information form will be filled in after meeting the pregnant women in the breathing exercise group admitted to the service at the first interview, giving information about the method to be followed in the practice, and obtaining their written consent. Since the hospitalization period of pregnant women hospitalized with the diagnosis of hyperemesis gravidarum varies between 3 and 7 days, the pregnant women with hyperemesis gravidarum who meet the research criteria are made 10 minutes once a day. A total of 1 times day diaphragmatic breathing exercise will be made on 3 consecutive days (5 minutes diaphragmatic breathing exercise, 5 minutes relaxation exercise). Diaphragmatic breathing exercises will be performed at least 4 hours after the use of antiemetic drugs in the service. Pre-test data will be obtained by using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales before the application. Afterward, 20 minutes from the application post-test data will be obtained by using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales. A total of 6 measurements will be made using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales before and after the diaphragmatic breathing exercises performed on the 1st, 2nd, and 3rd days.

Guided Imagery Group: An introductory information form will be filled in after meeting the pregnant women in the guided imagery group admitted to the service at the first interview, giving information about the method to be followed in the practice, and obtaining their written consent. 10 minutes once a day for pregnant women with hyperemesis gravidarum who meet the research criteria the guided imagery compact disc will be played with the computer. A guided imagery compact disc will be watched at least 4 hours after the use of antiemetic drugs in the service. Pre-test data will be obtained by using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales before the application. Afterward, 20 minutes from the application post-test data will be obtained by using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales. A total of 6 measurements will be made using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales before and after the guided imagery compact disc application on the 1st, 2nd, and 3rd days.

Control Group: No intervention will be made to the pregnant women in the control group, other than their routine daily care. Pre-test data will be obtained by applying the scales at least 4 hours after the use of antiemetic drugs in the service. 20 min from the pre-test data. Afterward, the final test data will be obtained by applying the scales. A total of 6 measurements will be made using the Nausea-Vomiting Severity Assessment Test in Pregnancy and Pregnancy-Related Anxiety Scale-R2 scales on the 1st, 2nd, and 3rd days.

2.5. Data Analysis: The data will analyze using Statistical Package for the Social Sciences 23.0 software. The analysis will be carried out by a statistician who was not included in the study. Tables will give frequency distribution (number, percentage) for categorical variables and descriptive statistics (median and quartiles, mean, standard deviation) for numerical variables. Shapiro Wilk test will use for conformity to the normal distribution and it will determine that numerical variables are not suitable for normal distribution. The Kruskal-Wallis test will use to determine whether there is a difference between the groups in terms of numerical measurements. In addition, Bonferroni correction will be applied while checking again with the Mann-Whitney U test from which group or groups the difference originated. The Chi-square test will be used to determine whether there is a difference between the groups in terms of categorical measures. Correlation (Spearman's rho) analysis will be conducted to see the direction and power of the correlation between variables. In comparison, the confidence interval will be taken as 95%, and the p significance level will accept as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and over,

  * Being primiparous,
  * Able to communicate verbally,
  * Agreeing to participate in the study,
  * Able to read and write,
  * 12th week of pregnancy and above
  * At least 3 days of hospitalization,
  * Having a single and live fetus,
  * No fetal congenital malformation,
  * Pregnant women who do not have systemic diseases (GIS, audiovestibular, endocrine, infection, and psychological) that may cause nausea and vomiting other than nausea and vomiting caused by pregnancy will be included in the study.

Exclusion Criteria:

* Having a risky pregnancy diagnosis;
* Obstetric complications,
* Having a psychiatric diagnosis,
* With systemic disease,

  * Having multiple pregnancies,
  * Fetal congenital malformation,
  * Pregnant women with systemic diseases that may cause nausea-vomiting will not be included in the study.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Nausea-Vomiting Severity | 20 minutes after interventions
  Nausea-Vomiting Severity Evaluation

SECONDARY OUTCOMES:
Pregnancy-Related Anxiety | 20 minutes after interventions
  Pregnancy-Related Anxiety Evaluation

CONTACTS AND LOCATIONS:
Overall Officials: EMİNE KARACAN, PhD, Study Director — ISKENDERUN TECHNICAL UNIVERSITY

REFERENCES:
- [Derived] Karacan E, Karacan E. Effects of guided imagery, and breathing exercise device on nausea-vomiting, and anxiety in hyperemesis gravidarum. J Reprod Infant Psychol. 2026 Jan 13:1-26. doi: 10.1080/02646838.2026.2615083. Online ahead of print. PMID 41531003